CLINICAL TRIAL: NCT03807778
Title: A Phase 1/2 Study of the Oral EGFR/HER2 Inhibitor TAK-788 in Japanese Non-Small Cell Lung Cancer Patients
Brief Title: A Study of Mobocertinib in Japanese Adults With Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-788-1003; U1111-1223-2659 (Other: WHO); jRCT2080224519 (Registry Identifier: jRCT)
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobocertinib, Phase 1 Part (Experimental): Mobocertinib 40 milligrams (mg) (as the starting dose), capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle for up to disease progression or intolerable toxicity, or another discontinuation criterion, and increasing until 160 mg, once daily (for up to approximately 10-12 cycles).
  Interventions: Drug: Mobocertinib
- Mobocertinib, Phase 2 Part (Experimental): Mobocertinib 160 mg, once daily, for up to approximately 10-12 cycles.
  Interventions: Drug: Mobocertinib

INTERVENTIONS:
Drug: Mobocertinib — Mobocertinib capsule.
  Other Names: TAK-788; AP32788

SUMMARY:
This study is in 2 parts. Different participants will take part in the 1st and 2nd parts of the study.

The main aim of the 1st part of the study is to check how much Mobocertinib adults with non-small cell lung cancer (NSCLC) can receive without getting side effects from it.

The main aim of the 2nd part of the study is to learn if the condition of adults with non-small cell lung cancer improves after treatment with Mobocertinib. Another aim is to continue checking for side effects from Mobocertinib.

In the 1st part of the study, at the first visit, the study doctor will check who can take part. For those that can take part, participants will take a capsule of Mobocertinib once a day for 28 days. This will count as 1 cycle. Different small groups of participants will receive lower to higher doses of Mobocertinib. The study doctors will check for side effects after each dose of TAK 788. In this way, researchers can work out the best dose of Mobocertinib to give participants in the 2nd part of the study.

Participants will visit the clinic 30 days after their treatment has finished for a final check-up.

In the 2nd part of the study, at the first visit, the study doctor will check who can take part. Participants will receive the best dose of Mobocertinib worked out from the 1st part of the study. Participants will receive Mobocertinib in the same way as those from the 1st part of the study. The study doctors will learn if the condition of these participants improves after treatment with Mobocertinib. The study doctors will also check for side effects from Mobocertinib.

After treatment has finished, participants will visit the clinic every 12 weeks until the end of the study.

In both parts of the study, participants can receive Mobocertinib for up to just over 1 year, or longer if their condition stays improved.

DETAILED DESCRIPTION:
The drug being tested in this study is called Mobocertinib. Mobocertinib is being tested to treat Japanese participants with NSCLC. This study has two parts (Phase 1 part and Phase 2 part), Phase 1 part of this study will look at the safety, efficacy, tolerability and PK of Mobocertinib orally administered once daily, and will determine a RP2D. Phase 2 study will look at the efficacy and safety of Mobocertinib in treatment naive Japanese NSCLC patients with epidermal growth factor receptor (EGFR) exon 20 insertion mutation. All participants will be assigned to Phase 1 part or Phase 2 part and will be asked to take Mobocertinib capsule as following dosage and regimen;

Phase 1 part; Mobocertinib, 40 mg as starting dose, once daily, and escalating up to 160 mg until a Maximum Tolerated Dose (MTD). An expansion phase may be followed at any dose to further confirm safety observations following identification of MTD/RP2D.

Phase 2 part; Mobocertinib, 160 mg, once daily

The study will enroll approximately 58-63 participants (Phase 1 part; 28-33 and Phase 2 part; 30).

This multi-center trial will be conducted in Japan. The overall time to participate in this study of Phase 1 part is approximately 3 years and Phase 2 part is approximately 4 years. Participants will make multiple visits to the clinic in the treatment period, and the post-treatment period including follow-up assessments after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria (Both in Phase 1 and Phase 2 Part);

1. Male or female patients ≥20 years old.
2. Must have measurable disease by RECIST v1.1. Previously irradiated lesions may not be used for target lesions, unless there is unambiguous radiological progression after radiotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
4. Minimum life expectancy of 3 months or more.
5. Adequate renal and hepatic function as defined by the following criteria:

   •Total serum bilirubin ≤1.5 × upper limit of normal (ULN) (≤3.0 × ULN for patients with Gilbert syndrome or if liver function abnormalities are due to underlying malignancy);

   •Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN (or ≤5 × ULN if liver function abnormalities are due to underlying malignancy);

   •Estimated creatinine clearance ≥30 mL/min (calculated by using the Cockcroft-Gault equation);

   •Serum albumin ≥2 g/dL; and

   •Serum lipase ≤1.5 × ULN; and

   •Serum amylase ≤1.5 × ULN unless the increased serum amylase is due to salivary isoenzymes.
6. Adequate bone marrow function as defined by the following criteria:

   * Absolute neutrophil count ≥1.5 × 109/L;
   * Platelet count ≥75 × 109/L in Phase 1 Part and ≥100 × 109/L in Phase 2 Part; and
   * Hemoglobin ≥9.0 g/dL.
7. Normal QT interval on screening ECG, defined as QTcF of ≤450 ms in males or ≤470 ms in females.
8. Female patients who:

   * Are postmenopausal (natural amenorrhea and not due to other medical reasons) for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective non-hormonal method of contraception and 1 additional effective (barrier) method (see Section 8.7.1) at the same time, from the time of signing the informed consent form (ICF) through 30 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.

Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.

Male patients, even if surgically sterilized (ie, status postvasectomy), who:

* Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study drug, OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject.

Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.

9.Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

10.Willingness and ability to comply with scheduled visits and study procedures.

* Phase-Specific Inclusion Criteria (Phase 1 part);

  1.Have histologically or cytologically confirmed locally advanced (and not a candidate for definitive therapy) (Stage IIIB) or metastatic NSCLC (Stage IV).

  2.Refractory to standard available therapies. 3.All toxicities from prior therapy have resolved to ≤ grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0), or have resolved to baseline, at the time of first dose of Mobocertinib. Note: treatment-related grade >1 alopecia or treatment-related grade 2 peripheral neuropathy are allowed if deemed irreversible.
* Phase-Specific Inclusion Criteria (Phase 2 part);

  1. Histologically or cytologically confirmed locally advanced not suitable for definitive therapy, recurrent, or metastatic (Stage IV) NSCLC.
  2. Not received prior systemic treatment for locally advanced or metastatic disease (with the exception below): Neoadjuvant or adjuvant chemotherapy/immunotherapy for Stage I to III or combined modality chemotherapy/radiation for locally advanced disease is allowed if completed >6 months before the development of metastatic disease.
  3. A documented EGFR in-frame exon 20 insertion (including A763_Y764insFQEA, V769_D770insASV, D770_N771insNPG, D770_N771insSVD, H773_V774insNPH, or any other in-frame exon 20 insertion mutation) by a local test that has been analytically validated per local authority guidelines. The EGFR exon 20 insertion mutation can be either alone or in combination with other EGFR or HER2 mutations except EGFR common mutations (exon 19 del or L858R).
  4. Adequate tumor tissue available, either from primary or metastatic sites, for central laboratory confirmation of EGFR in-frame exon 20 insertion mutation. Note: confirmation of central test positivity is not required before the first dose of Mobocertinib.

     Exclusion Criteria:

     General Exclusion Criteria (Both in Phase 1 and Phase 2 Part);

  <!-- -->

  1. Have been diagnosed with another primary malignancy other than NSCLC except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
  2. Have undergone major surgery within 28 days prior to first dose of Mobocertinib. Minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
  3. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic).
  4. Have significant, uncontrolled, or active cardiovascular disease, including, but not restricted to:
* Myocardial infarction within 6 months prior to the first dose of study drug;
* Unstable angina within 6 months prior to first dose;
* Congestive heart failure within 6 months prior to first dose;
* History of clinically significant (as determined by the treating physician) atrial arrhythmia;
* Any history of ventricular arrhythmia; or
* Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose.

  5.Have uncontrolled hypertension. Patients with hypertension should be under treatment on study entry to control blood pressure.

  6.Currently being treated with medications known to be associated with the development of Torsades de Pointes.

  7.Have an ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics. Have a known history of HIV infection. Testing of HIV is not required in the absence of history.Hepatitis B surface antigen (HBsAg) positive patients are allowed to enroll if hepatitis B virus (HBV)-DNA is below 1000 copies/mL in the plasma.Patients who have positive hepatitis C virus (HCV) antibody can be enrolled but must have HCV-RNA undetectable in the plasma.

  8.Currently have or have a history of interstitial lung disease (ILD), radiation pneumonitis that required steroid treatment, or drug-related pneumonitis.

  9.Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period.
* Note: Female patients who are lactating will be eligible if they discontinue breastfeeding.

  10.Have gastrointestinal illness or disorder that could affect oral absorption of Mobocertinib.

  11.Have any condition or illness that, in the opinion of the investigator, might compromise patient safety or interfere with the evaluation of the safety of the drug.
* Phase-Specific Exclusion Criteria (Phase 1 part);

  1. Previously received Mobocertinib.
  2. Received small-molecule anticancer therapy (including cytotoxic chemotherapy and investigational agents) within 14 days prior to the first dose of Mobocertinib (except for reversible EGFR TKIs [ie, erlotinib or gefitinib] up to 7 days prior to the first dose of Mobocertinib).
  3. Received antineoplastic monoclonal antibodies including immunotherapy within 28 days prior to the first dose of Mobocertinib.
  4. Received radiotherapy within 14 days prior to the first dose of Mobocertinib, Stereotactic radiosurgery (SRS) and stereotactic body radiosurgery are allowed up to 7 days prior to the first dose.
  5. Have symptomatic CNS metastases (parenchymal or leptomeningeal) at screening or asymptomatic disease requiring corticosteroids to control symptoms within 7 days prior to the first dose of Mobocertinib.

     Note: If a patient has worsening neurological symptoms or signs due to CNS metastases, the patient needs to complete local therapy and be neurologically stable (with no requirement for corticosteroids or use of anticonvulsants) for 7 days prior to the first dose of Mobocertinib. Patients with no prior history of signs or symptoms of CNS metastases but who receive prophylactic steroids or anticonvulsants are allowed.
  6. Received a strong cytochrome P450 (CYP)3A inhibitor or strong CYP3A inducer within 2 weeks prior to first dose of Mobocertinib.
* Phase-Specific Exclusion Criteria (Phase 2 part);

  1. Received radiotherapy within 14 days before the first dose of Mobocertinib or has not recovered from radiotherapy-related toxicities. Stereotactic radiosurgery, stereotactic body radiotherapy, or palliative radiation outside the chest and brain is allowed up to 7 days before the first dose of Mobocertinib.
  2. Have known active brain metastases (have either previously untreated intracranial CNS metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions). Brain metastases are allowed if they have been treated with surgery and/or radiation and have been stable without requiring corticosteroids to control symptoms within 7 days before the first dose of Mobocertinib, and have no evidence of new or enlarging brain metastases.
  3. Received a moderate or strong CYP3A inhibitor or moderate or strong CYP3A inducer within 10 days prior to first dose of Mobocertinib.
  4. Have cardiac ejection fraction <50% by echocardiogram or multigated acquisition (MUGA) scan at screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- Japan (25):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Cente, Akashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Okayama University Hospital, Kita-ku, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Cancer Center, Shinden, Saitama
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - Yamaguchi Ube Medical Center, Ube, Yamaguchi
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Tokushima University Hospital, Tokushima
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Yang JC, Zhou C, Janne PA, Ramalingam SS, Kim TM, Riely GJ, Spira AI, Piotrowska Z, Mekhail T, Garcia Campelo MR, Felip E, Bazhenova L, Jin S, Kaur M, Diderichsen PM, Gupta N, Bunn V, Lin J, N Churchill E, Mehta M, Nguyen D. Characterization and management of adverse events observed with mobocertinib (TAK-788) treatment for EGFR exon 20 insertion-positive non-small cell lung cancer. Expert Rev Anticancer Ther. 2023 Jan;23(1):95-106. doi: 10.1080/14737140.2023.2157815. Epub 2022 Dec 28. PMID 36537204
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a2bd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites for Phase 1 and 17 investigative sites for Phase 2 in Japan from 04 February 2019. The study is currently ongoing. Results in this summary are reported based on the primary completion date (08 November 2021) of the study.
Pre-assignment Details: Participants with a diagnosis of locally advanced or metastatic non-small cell lung cancer (NSCLC) were enrolled in a Dose Escalation Phase 1 Part of the study to receive mobocertinib (40, 120 or 160 milligram [mg]) and participants with locally advanced or metastatic NSCLC harboring epidermal growth factor receptor (EGFR) exon 20 insertion mutations were enrolled in Phase 2 Part of the study to receive RP2D of mobocertinib confirmed from the Phase 1 Part.
Groups:
- Mobocertinib 40 mg, Phase 1 Part: Mobocertinib 40 mg (as the starting dose), capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC.
- Mobocertinib 120 mg, Phase 1 Part: Mobocertinib 120 mg, capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC.
- Mobocertinib 160 mg, Phase 1 Part: Mobocertinib 160 mg, capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC.
- Mobocertinib 160 mg, Phase 2 Part: Mobocertinib 160 mg, capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC harboring EGFR exon 20 insertion mutations.
Period: Overall Study
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 2 Part
Started | 4 | 4 | 12 | 33
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 12 | 33
Not completed — Adverse Event | 0 | 0 | 3 | 5
Not completed — Progressive Disease | 4 | 2 | 8 | 15
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Ongoing at data cut- off date (08 November 2021) | 0 | 0 | 1 | 11

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of mobocertinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 2 Part | Total
Number analyzed (Participants) | 4 | 4 | 12 | 33 | 53
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 50 | 1 | 1 | 2 | 4 | 8
  Greater than or equal to (>=) 50 to < 65 years | 1 | 1 | 4 | 12 | 18
  >=65 to <75 years | 2 | 2 | 5 | 11 | 20
  >=75 years | 0 | 0 | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 9 | 21 | 35
  Male | 2 | 1 | 3 | 12 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 12 | 33 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 4 | 12 | 33 | 53
Disease Stage at Screening [Count of Participants; unit: Participants] — Cancer stage is a measure of disease progression. The later stage indicates more advanced cancer. So, the Participants with Stage IV cancer had more advanced disease than stage III participants. The letters represent sub groups within a given stage, with B representing more advanced cancer than A. Other: Unknown or not staged.
  Participants
    IIIB | 0 | 0 | 1 | 0 | 1
    IV | 4 | 4 | 11 | 0 | 19
    IVA | 0 | 0 | 0 | 16 | 16
    IVB | 0 | 0 | 0 | 15 | 15
    Other | 0 | 0 | 0 | 2 | 2
Time Since Initial Diagnosis [Median (Full Range); unit: months] | 26.90 [17.9 to 157.8] | 15.50 [11.8 to 31.6] | 20.20 [2.6 to 100.4] | 1.90 [0.5 to 166.0] | 9.4 [0.5 to 166.0]
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG-PS assessed participant's performance status scale of 0 to 5: 0=Fully active/able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (> [greater than] 50% of waking hours), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. A higher score indicated greater functional impairment.
  Participants
    0 | 2 | 0 | 5 | 21 | 28
    1 | 2 | 4 | 7 | 12 | 25
Central Nervous System (CNS) involvement at Screening [Count of Participants; unit: Participants]
  Was involved | 2 | 4 | 4 | 16 | 26
  Was not involved | 2 | 0 | 8 | 17 | 27
Histopathological Classification of NSCLC [Count of Participants; unit: Participants] — Participants with NSCLC were categorized into adenocarcinoma, adenosquamous carcinoma, large cell, squamous, unknown and other.
  Participants
    Adenocarcinoma | 4 | 4 | 12 | 33 | 53
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 2 | 2 | 8 | 17 | 29
  Former Smoker | 2 | 2 | 4 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Part: Recommended Phase 2 Dose (RP2D) of Orally Administered Mobocertinib
Description: The RP2D was the maximum tolerated dose (MTD) or less. The MTD was declared when at least 9 participants were evaluable in the study and 6 participants were evaluable at the current dose, and the current dose was recommended for the next cohort. The dose recommended for use in phase 2 part was analyzed on the basis of the safety and tolerability data obtained in phase 1 part of the study.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: The dose-limiting toxicity (DLT)-evaluable population included all participants who received at least 75 percent (%) of their planned mobocertinib doses for their first cycle of treatment (unless interrupted by study drug-related AEs). As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Number; unit: mg
Groups:
- Mobocertinib, Phase 1 Part: All Participants: Mobocertinib 40, 120 or 160 mg capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC.
Arm/Group | Mobocertinib, Phase 1 Part: All Participants
Number analyzed (Participants) | 16
mg | 160

2. Primary Outcome: Phase 2 Part: Confirmed Objective Response Rate (ORR) as Assessed by the Independent Review Committee (IRC)
Description: Confirmed ORR is defined as percentage of participants who were confirmed to had achieved complete response (CR) or partial response (PR) per IRC using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment. Confirmed responses were responses that persisted on repeat imaging >=4 weeks after initial response. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 millimeter (mm) in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR (target lesions): at least 30% decrease in sum of the longest diameters (SLD) of target lesions, taking as reference baseline sum diameters. The SLD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the first dose of the study drug until progressive disease (PD) (up to 2 years and 9 months)
Population: The centrally confirmed population was defined as the participants who had confirmed harboring EGFR exon 20 insertion mutation by central test and had received at least 1 dose of mobocertinib. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure. As planned, this outcome measure was assessed only for Phase 2 Part of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 14
percentage of participants | 28.6 [10.4 to 54.0]

3. Secondary Outcome: Phase 1 Part: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: From first dose of study drug until 30 days after the last dose or before initiation of new anticancer therapy (whichever comes first) (Up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: The safety population included all participants who received at least 1 dose of mobocertinib. As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 12
Participants | 3 | 4 | 12

4. Secondary Outcome: Phase 1 Part: Number of Participants With First Cycle DLTs Based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.00
Description: DLT was defined as drug-related toxicity which met one of the following criteria and occurred within the first 28 days of study treatment (Cycle 1): Non-hematologic toxicities any >=grade (G) 3 non-hematologic toxicity, with exception of self-limiting or medically controllable toxicities(nausea, vomiting, fatigue, electrolyte disturbances, hypersensitivity reactions) lasting <3 days, excluding alopecia. Hematologic toxicities: febrile neutropenia not related to underlying disease (fever,>38.3 degree Celsius [C]); absolute neutrophil count <0.5*10^9 per liter [/L]); prolonged G4 neutropenia (>=7 days) (if granulocyte-colony stimulating factor [G-CSF] required, event considered as DLT irrespective of the duration); neutropenic infection:>=G3 neutropenia with >=G3 infection; thrombocytopenia >=G3 with bleeding, >=G3 requiring platelet transfusion or G4 without bleeding lasting >=7 days. Missed >=25% of planned doses of drug over 28 days due to treatment-related AEs in first cycle.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: The DLT-evaluable population included as all participants who received at least 75% of their planned mobocertinib doses for their first cycle of treatment (unless interrupted by study drug-related AEs). As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 8
Participants | 0 | 1 | 2

5. Secondary Outcome: Phase 1 Part: Number of DLTs for Mobocertinib Based on NCI CTCAE, Version 5.00
Description: DLT was defined as drug-related toxicity which met one of the following criteria and occurred within the first 28 days of study treatment (Cycle 1): Non-hematologic toxicities any >=G 3 non-hematologic toxicity, with exception of self-limiting or medically controllable toxicities (nausea, vomiting, fatigue, electrolyte disturbances, hypersensitivity reactions) lasting <3 days, excluding alopecia. Hematologic toxicities: febrile neutropenia not related to underlying disease (fever,>38.3 degree C); absolute neutrophil count <0.5*10^9/L); prolonged G4 neutropenia (>=7 days) (if granulocyte-colony stimulating factor [G-CSF] required, event considered as DLT irrespective of the duration); neutropenic infection: >=G3 neutropenia with >=G3 infection; thrombocytopenia >=G3 with bleeding, >=G3 requiring platelet transfusion or G4 without bleeding lasting >=7 days. Missed >=25% of planned doses of drug over 28 days due to treatment-related AEs in first cycle.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: as for outcome 4
Measure: Number; unit: DLTs
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 8
DLTs | 0 | 1 | 4

6. Secondary Outcome: Phase 1 Part: Maximum Tolerated Dose (MTD) of Orally Administered Mobocertinib
Description: The MTD was declared when at least 9 participants were evaluable in the study and 6 participants were evaluable at the current dose, and the current dose was recommended for the next cohort.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: The DLT-evaluable population was defined as all participants who received at least 75% of their planned mobocertinib doses for their first cycle of treatment (unless interrupted by study drug-related AEs). As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Number; unit: mg
Arm/Group | Mobocertinib, Phase 1 Part: All Participants
Number analyzed (Participants) | 16
mg | 160

7. Secondary Outcome: Phase 1 Part, Cmax: Maximum Observed Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) After a Single Oral Dose
Time Frame: Cycle 1 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: The pharmacokinetic (PK) population included all participants for whom there were sufficient dosing and mobocertinib concentration-time data to reliably estimate the PK parameters. As planned, this outcome measure was assessed only for Phase 1 Part of the study
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 12
nanogram per milliliter (ng/mL)
  Mobocertinib | 15.40 (76.1) | 70.28 (56.2) | 100.2 (36.3)
  AP32960 | 8.797 (96.4) | 28.81 (31.0) | 47.84 (28.9)
  AP32914 | 1.677 (66.2) | 4.962 (41.7) | 8.626 (40.6)

8. Secondary Outcome: Phase 1 Part, Tmax: Time of First Occurrence of Cmax for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) After a Single Oral Dose
Time Frame: Cycle 1 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: The PK population included all participants for whom there were sufficient dosing and mobocertinib concentration-time data to reliably estimate the PK parameters. As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Median (Full Range); unit: hour
Groups:
- Mobocertinib 120 mg, Phase 1 Part: Mobocertinib 120 mg, capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle disease until progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC.
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 12
hour
  Mobocertinib | 3.830 [3.83 to 3.88] | 3.985 [3.88 to 5.92] | 3.985 [3.83 to 7.87]
  AP32960 | 3.830 [3.83 to 5.88] | 3.985 [3.88 to 5.92] | 4.965 [3.83 to 7.87]
  AP32914 | 3.830 [3.83 to 5.88] | 4.995 [3.88 to 5.98] | 4.965 [3.83 to 7.87]

9. Secondary Outcome: Phase 1 Part, AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) After a Single Oral Dose
Time Frame: Cycle 1 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: The PK population included all participants for whom there were sufficient dosing and mobocertinib concentration-time data to reliably estimate the PK parameters. Here number analyzed 'n' signifies participants who were evaluable for specified categories. As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 4 | 4 | 12
hour*nanogram per milliliter (h*ng/mL)
  Mobocertinib | 152.9 (62.2) | 858.1 (60.3) | 1196 (43.0)
  AP32960 | 86.06 (77.2) | 378.2 (35.3) | 569.9 (27.1)
  AP32914: number analyzed (Participants) | 3 | 4 | 12
  AP32914 | 20.15 (39.6) | 70.58 (45.6) | 105.9 (44.5)

10. Secondary Outcome: Phase 1 Part, Cmax, ss: Maximum Observed Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) at Steady State After Multiple Oral Doses
Time Frame: Cycle 2 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: The PK population included all participants for whom there were sufficient dosing and mobocertinib concentration-time data to reliably estimate the PK parameters. Here overall number of participants analyzed signifies participants who were evaluable for this outcome measure. As planned, this outcome measure was assessed only for Phase 1 Part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 3 | 2 | 5
ng/mL
  Mobocertinib | 17.90 (34.4) | 106.2 (39.4) | 90.00 (18.4)
  AP32960 | 12.34 (68.7) | 59.94 (24.3) | 56.85 (21.0)
  AP32914 | 1.808 (31.4) | 9.198 (37.7) | 7.920 (13.3)

11. Secondary Outcome: Phase 1 Part, Tmax, ss: Time of First Occurrence of Cmax for Mobocertinib Its Active Metabolites (AP32960 and AP32914) at Steady State After Multiple Oral Doses
Time Frame: Cycle 2 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 3 | 2 | 5
hour
  Mobocertinib | 3.950 [3.83 to 4.05] | 4.000 [3.97 to 4.03] | 3.970 [3.92 to 5.95]
  AP32960 | 3.950 [3.83 to 4.05] | 4.000 [3.97 to 4.03] | 3.970 [3.92 to 5.95]
  AP32914 | 3.950 [3.83 to 4.05] | 4.000 [3.97 to 4.03] | 3.980 [3.92 to 5.95]

12. Secondary Outcome: Phase 1 Part, AUC24, ss: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) at Steady State After Multiple Oral Doses
Time Frame: Cycle 2 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 3 | 2 | 5
h*ng/mL
  Mobocertinib | 214.8 (29.9) | 1195 (50.1) | 1141 (25.9)
  AP32960 | 158.6 (63.1) | 794.0 (36.6) | 750.3 (27.4)
  AP32914 | 21.02 (24.3) | 116.9 (49.7) | 105.0 (20.4)

13. Secondary Outcome: Phase 1 Part, Rac (AUC 24): Extent of Accumulation Ratio Based on AUC 24 on Multiple Dosing for Mobocertinib and Its Active Metabolites (AP32960 and AP32914) at Steady State After Multiple Oral Doses
Description: Rac (AUC 24) was calculated as the ratio of drug concentrations observed during a dosing interval at steady state divided by drug concentrations seen during the dosing interval after a single (first) dose. Rac (AUC 24) = AUC(0-24) on Cycle 2 Day 1/ AUC(0-24) on Cycle 1 Day 1.
Time Frame: Cycle 2 Day 1: pre-dose and at 0.5 1, 2, 4, 6, 8 and 24 hours post-dose (Cycle length = 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 3 | 2 | 5
ratio
  Mobocertinib | 1.096 (43.8) | 1.260 (12.9) | 0.9227 (39.3)
  AP32960 | 1.393 (17.5) | 1.765 (2.0) | 1.366 (15.9)
  AP32914 | 1.044 (41.7) | 1.414 (21.2) | 1.027 (34.5)

14. Secondary Outcome: Phase 1 Part: ORR in Participants With EGFR Mutations as Assessed by Investigator
Description: Investigator assessed ORR using RECIST version 1.1 in participants with EGFR mutations. ORR was defined as the percentage of participants achieving CR and PR per RECIST version 1.1. Confirmed responses were responses that persisted on repeat imaging >=4 weeks after initial response. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR (target lesions): at least 30% decrease in SLD of target lesions, taking as reference baseline sum diameters. All participants with ORR had documentation of EGFR exon 20 insertion mutation.
Time Frame: From the first dose of the study drug until PD (up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: The response-evaluable population was defined as participants who received at least 1 dose of mobocertinib, had measurable disease at baseline, and at least 1 post-baseline response assessment. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure. As planned, this outcome measure was assessed only for Phase 1 Part of study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 3 | 4 | 11
percentage of participants | 0.0 [0.000 to 70.760] | 25.0 [0.631 to 80.588] | 18.2 [2.283 to 51.776]

15. Secondary Outcome: Phase 1 Part: ORR in Participants With HER2 Mutations as Assessed by Investigator
Description: Investigator assessed ORR using RECIST version 1.1 in participants with HER2 mutations. ORR was defined as the percentage of participants achieving CR and PR per RECIST version 1.1. Confirmed responses were responses that persisted on repeat imaging >=4 weeks after initial response. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR (target lesions): at least 30% decrease in SLD of target lesions, taking as reference baseline sum diameters.
Time Frame: From the first dose of the study drug until PD (up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part
Number analyzed (Participants) | 1 | 0 | 0
percentage of participants | 0 [0.000 to 97.500] |  |

16. Secondary Outcome: Phase 2 Part: Confirmed ORR as Assessed by the Investigator
Description: Confirmed ORR was defined as the percentage of the participants who were confirmed to have achieved CR or PR per the investigator using RECIST version 1.1. Confirmed responses were responses that persisted on repeat imaging >=4 weeks after initial response. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR (target lesions): at least 30% decrease in SLD of target lesions, taking as reference baseline sum diameters.
Time Frame: From the first dose of the study drug until PD (up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: The centrally confirmed population was defined as the participants who had confirmed harboring EGFR exon 20 insertion mutation by central test and had received at least 1 dose of mobocertinib. As planned, this outcome measure was assessed only for Phase 2 Part of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
percentage of participants | 43.5 [23.2 to 65.5]

17. Secondary Outcome: Phase 2 Part: Duration of Response (DOR) as Assessed by the IRC as Per RECIST V1.1
Description: Duration of response as assessed by the IRC was defined as the time interval from first documentation of CR/PR (whichever is first recorded) until the first date that PD is objectively documented. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level; PR: At least a 30% decrease in SLD of target lesions, taking as a reference the baseline SLD. PD (target lesion response): SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest); PD (non-target lesion response): Unequivocal progression of existing non-target lesions. The SLD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first documentation of CR/PR until first PD (Up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 3
months | 7.4 [7.3 to NA] — Upper limit of 95% confidence interval (CI) was not reached due to low number of participants with events.

18. Secondary Outcome: Phase 2 Part: DOR as Assessed by Investigator as Per RECIST V1.1
Description: Duration of response as assessed by the investigator was defined as the time interval from first documentation of CR/PR (whichever is first recorded) until the first date that PD is objectively documented. CR (target lesion response):disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level; PR: At least a 30% decrease in SLD of target lesions, taking as a reference the baseline SLD. PD (target lesion response): SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest); PD (non-target lesion response): Unequivocal progression of existing non-target lesions. The SLD must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first documentation of CR/PR until first PD (Up to 2 years and 9 months, till data cut-off of 08 November 2021)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 10
months | 6.6 [1.8 to NA] — Upper limit of 95% CI was not reached due to low number of participants with events.

19. Secondary Outcome: Phase 2 Part: Time to Response as Assessed by the IRC as Per RECIST V1.1
Description: Time to response as assessed by the IRC was defined as the time interval from the date of the first dose of study treatment until the initial observation of CR or PR for participants with confirmed CR/PR. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose of the study drug up to first confirmed CR or PR (Up to 2 years 9 months, till data cut-off of 08 November 2021)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 3
days | 52.0 [51 to 58]

20. Secondary Outcome: Phase 2 Part: Time to Response as Assessed by the Investigator Per RECIST V1.1
Description: Time to response as assessed by the investigator was defined as the time interval from the date of the first dose of study treatment until the initial observation of CR or PR for participants with confirmed CR/PR. CR (target lesion response): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion response): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 10
days | 57.0 [52 to 168]

21. Secondary Outcome: Phase 2 Part: Disease Control Rate (DCR) as Assessed by the IRC as Per RECIST V1.1
Description: DCR as assessed by IRC was defined as percentage of participants achieved CR, PR, stable disease (SD) (measurements must had met SD criteria at least once after study entry at minimum interval of 42 days) after initiation of study drug.CR(target lesion): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis.CR(non-target lesion): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level.PR(target lesions): at least 30% decrease in SLD of target lesions, taking as reference baseline sum diameters.SD(target lesion): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.PD(target lesion): SLD increased by at least 20% from smallest value on study, SLD must also demonstrate an absolute increase of at least 5 mm.PD (non-target lesion): unequivocal progression of existing non-target lesions.
Time Frame: From the first dose of the study drug until PD (Up to 2 years 9 month, till data cut-off of 08 November 2021)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
percentage of participants | 82.6 [61.2 to 95.0]

22. Secondary Outcome: Phase 2 Part: DCR as Assessed by the Investigator Per RECIST V1.1
Description: DCR as assessed by investigator was defined as percentage of participants achieved CR, PR, SD (measurements must had met SD criteria at least once after study entry at minimum interval of 42 days) after initiation of study drug. CR (target lesion): disappearance of all extranodal target lesions, all pathological lymph nodes must have decreased to <10 mm in short axis. CR (non-target lesion): disappearance of all extranodal nontarget lesions, all lymph nodes must be nonpathological in size (<10 mm short axis) and normalization of tumor marker level. PR (target lesions): at least 30% decrease in SLD of target lesions, taking as reference baseline sum diameters.SD (target lesion): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD(target lesion): SLD increased by at least 20% from smallest value on study, SLD must also demonstrate an absolute increase of at least 5 mm.PD (non-target lesion): unequivocal progression of existing non-target lesions.
Time Frame: From the first dose of the study drug until PD (Up to 2 years 9 month, till data cut-off of 08 November 2021)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
percentage of participants | 91.3 [72.0 to 98.9]

23. Secondary Outcome: Phase 2 Part: Progression Free Survival (PFS) as Assessed by the IRC as Per RECIST V1.1
Description: PFS as assessed by the IRC was defined as the time interval from the start of study treatment until to the first documentation of PD or death due to any cause (whichever comes first) according to RECIST version 1.1.PD (target lesion response): SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest). The SLD must also demonstrate an absolute increase of at least 5 mm. PD (non-target lesion response): unequivocal progression of existing non-target lesions.
Time Frame: From the first dose of the study drug until PD or death due to any cause (whichever comes first) (Up to 2 years and 9 months, till data cut-off of 08 November 2021
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Mobocertinib 160 mg, Phase 2 Part: Mobocertinib 160 mg, capsules, orally, once daily on Days 1-28 of each 28-day treatment cycle until disease progression or intolerable toxicity, or another discontinuation criterion in participants with locally advanced or metastatic NSCLC harboring EGFR exon 20 insertion mutations in participants with locally advanced or metastatic NSCLC harboring EGFR exon 20 insertion mutations.
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
months | 9.3 [7.4 to NA] — Upper limit of 95% CI was not reached due to low number of participants with events.

24. Secondary Outcome: Phase 2 Part: PFS as Assessed by the Investigator as Per RECIST V1.1
Description: PFS as assessed by the investigator was defined as the time interval from the start of study treatment until to the first documentation of PD or death due to any cause (whichever comes first) according to RECIST version 1.1.PD (target lesion response): SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest). The SLD must also demonstrate an absolute increase of at least 5 mm. PD (non-target lesion response): unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 23
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
months | 9.2 [6.2 to NA] — Upper limit of 95% CI was not reached due to low number of participants with events.

25. Secondary Outcome: Phase 2 Part: Overall Survival (OS)
Description: OS was defined as the interval from the date of the first dose of the study treatment until death due to any cause.
Time Frame: From the start of the study drug up to death due to any cause (Up to 2 years 9 months, till data cut-off of 08 November 2021)
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 23
months | NA [NA to NA] — Median, lower and upper limit of 95% CI were not reached due to low number of participants with events.

26. Secondary Outcome: Phase 2 Part: Change From Baseline in Patient-reported Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30
Description: EORTC QLQ-C30, version 3.0 was a cancer-specific questionnaire comprised of 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); a global health status (GHS)/quality-of-life (QoL) scale; and a six single-item scales (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). Raw scores converted into scale scores ranging from 0 to 100. For functional and GHS/QoL scales, higher scores represent better HRQoL (positive change from Baseline=improvement), for symptom scales lower scores represent better QoL (i.e., a low level of symptomatology/problems) (negative change from Baseline=improvement), and for six-single item scale, lower scores represent better HRQoL (negative change from Baseline=improvement).
Time Frame: Baseline and at 30 days after last dose (at Month 19)
Population: FAS included all participants who received at least one dose of mobocertinib. Here number analyzed 'n' signifies participants who were evaluable for specified categories. As planned, this outcome measure was assessed only for Phase 2 Part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 33
score on a scale
  Global Health Status: Baseline | 64.7 (18.79)
  Global Health Status: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Global Health Status: Change from Baseline at 30 Days After Last Dose | -4.0 (17.45)
  Physical Functioning: Baseline | 85.5 (14.03)
  Physical Functioning: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Physical Functioning: Change from Baseline at 30 Days After Last Dose | -34.6 (40.38)
  Role Functioning: Baseline | 80.3 (25.78)
  Role Functioning: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Role Functioning: Change from Baseline at 30 Days After Last Dose | -53.4 (50.57)
  Emotional Functioning: Baseline | 80.8 (20.13)
  Emotional Functioning: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Emotional Functioning: Change from Baseline at 30 Days After Last Dose | -6.0 (12.00)
  Cognitive Functioning: Baseline | 84.2 (16.09)
  Cognitive Functioning: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Cognitive Functioning: Change from Baseline at 30 Days After Last Dose | 4.3 (8.50)
  Social Functioning: Baseline | 87.4 (18.54)
  Social Functioning: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Social Functioning: Change from Baseline at 30 Days After Last Dose | -12.5 (15.84)
  Fatigue: Baseline | 27.8 (20.85)
  Fatigue: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Fatigue: Change from Baseline at 30 Days After Last Dose | 29.0 (38.28)
  Nausea and Vomiting: Baseline | 3.6 (12.42)
  Nausea and Vomiting: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Nausea and Vomiting: Change from Baseline at 30 Days After Last Dose | 0.0 (12.02)
  Pain: Baseline | 19.2 (21.21)
  Pain: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Pain: Change from Baseline at 30 Days After Last Dose | 9.6 (18.90)
  Dyspnoea: Baseline | 23.1 (26.94)
  Dyspnoea: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Dyspnoea: Change from Baseline at 30 Days After Last Dose | 13.6 (38.11)
  Insomnia: Baseline | 26.2 (24.72)
  Insomnia: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Insomnia: Change from Baseline at 30 Days After Last Dose | 20.2 (50.51)
  Appetite Loss: Baseline | 22.1 (25.91)
  Appetite Loss: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Appetite Loss: Change from Baseline at 30 Days After Last Dose | 20.2 (30.02)
  Constipation: Baseline | 14.1 (23.56)
  Constipation: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 5
  Constipation: Change from Baseline at 30 Days After Last Dose | -6.8 (27.85)
  Diarrhoea: Baseline | 6.0 (15.46)
  Diarrhoea: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Diarrhoea: Change from Baseline at 30 Days After Last Dose | -8.3 (31.60)
  Financial Difficulties: Baseline | 9.0 (14.92)
  Financial Difficulties: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Financial Difficulties: Change from Baseline at 30 Days After Last Dose | 8.3 (16.50)

27. Secondary Outcome: Phase 2 Part: Change From Baseline in Patient-reported Symptoms (Particular Core Symptoms of Lung Cancer), Functioning, and HRQoL as Assessed by the EORTC Lung Cancer Module QLQ-LC13
Description: HRQOL scores was assessed with EORTC, it is a lung cancer module QLQ-LC13, version 3.0. QLQ-LC13 included 13 questions (4-point scale where 1=Not at all [best] to 4=Very much [worst]) assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain [chest, arm or shoulder, other parts]), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Subscale score range: 0 to 100. Higher symptom score = greater degree of symptom severity.
Time Frame: Baseline and at 30 days after last dose (at Month 19)
Population: The full analysis set (FAS) included all participants who received at least one dose of mobocertinib. Here number analyzed 'n' signifies participants who were evaluable for specified categories. As planned, this outcome measure was assessed only for Phase 2 Part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobocertinib 160 mg, Phase 2 Part
Number analyzed (Participants) | 33
score on a scale
  Dyspnoea: Baseline | 16.4 (15.76)
  Dyspnoea: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Dyspnoea: Change from Baseline at 30 Days After Last Dose | 2.8 (18.79)
  Coughing: Baseline | 27.1 (24.24)
  Coughing: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Coughing: Change from Baseline at 30 Days After Last Dose | -8.5 (41.99)
  Haemoptysis: Baseline | 2.0 (8.00)
  Haemoptysis: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Haemoptysis: Change from Baseline at 30 Days After Last Dose | 0.0 (0.0)
  Sore Mouth: Baseline | 5.0 (12.02)
  Sore Mouth: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Sore Mouth: Change from Baseline at 30 Days After Last Dose | 0.0 (0.0)
  Dysphagia: Baseline | 7.0 (13.70)
  Dysphagia: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Dysphagia: Change from Baseline at 30 Days After Last Dose | 0.0 (0.0)
  Peripheral Neuropathy: Baseline | 6.0 (15.46)
  Peripheral Neuropathy: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Peripheral Neuropathy: Change from Baseline at 30 Days After Last Dose | -8.3 (16.50)
  Alopecia: Baseline | 9.0 (20.80)
  Alopecia: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Alopecia: Change from Baseline at 30 Days After Last Dose | 0.0 (0.0)
  Pain in Chest: Baseline | 14.1 (20.42)
  Pain in Chest: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Pain in Chest: Change from Baseline at 30 Days After Last Dose | -8.3 (16.50)
  Pain in Arm or Shoulder: Baseline | 17.0 (18.75)
  Pain in Arm or Shoulder: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Pain in Arm or Shoulder: Change from Baseline at 30 Days After Last Dose | -8.3 (16.50)
  Pain in Other Parts: Baseline | 18.1 (22.17)
  Pain in Other Parts: Change from Baseline at 30 Days After Last Dose: number analyzed (Participants) | 4
  Pain in Other Parts: Change from Baseline at 30 Days After Last Dose | -8.3 (16.50)

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after the first dose of study drug up to 30 days after the last dose of study drug or initiation of the subsequent anticancer therapies, whichever comes first (Up to 2 years and 9 months, till data cut-off of 08 November 2021)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Mobocertinib 40 mg, Phase 1 Part | Mobocertinib 120 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 1 Part | Mobocertinib 160 mg, Phase 2 Part
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 0/12 | 2/33
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/4 | 3/12 | 11/33
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 12/12 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobocertinib 40 mg, Phase 1 Part (N=4) | Mobocertinib 120 mg, Phase 1 Part (N=4) | Mobocertinib 160 mg, Phase 1 Part (N=12) | Mobocertinib 160 mg, Phase 2 Part (N=33)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mobocertinib 40 mg, Phase 1 Part (N=4) | Mobocertinib 120 mg, Phase 1 Part (N=4) | Mobocertinib 160 mg, Phase 1 Part (N=12) | Mobocertinib 160 mg, Phase 2 Part (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 12 | 33
Nausea (Gastrointestinal disorders) | 2 | 2 | 7 | 19
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 8 | 21
Vomiting (Gastrointestinal disorders) | 0 | 2 | 7 | 7
Angular cheilitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 4 | 4
Malaise (General disorders) | 0 | 1 | 1 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Paronychia (Infections and infestations) | 0 | 1 | 6 | 21
Hordeolum (Infections and infestations) | 0 | 0 | 2 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 5 | 8
Blood creatinine increased (Investigations) | 0 | 0 | 5 | 8
Lymphocyte count decreased (Investigations) | 0 | 1 | 4 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 5
Lipase increased (Investigations) | 0 | 1 | 3 | 12
Weight decreased (Investigations) | 0 | 1 | 2 | 13
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4 | 9
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 3 | 6
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 3
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 8 | 13
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 7 | 14
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 14
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 3 | 4
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03807778/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03807778/SAP_001.pdf